CLINICAL TRIAL: NCT02119884
Title: Hemodynamic Effects of Terlipressin and High Dose Octreotide on Patients With Liver Cirrhosis Related Esophageal Varices: A Randomized, Placebo-controlled Multicenter Trial
Brief Title: Hemodynamic Effects of Terlipressin and High Dose Octreotide
Acronym: HEofT&O
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Shandong Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Shiyao Chen, department of Gastroenterology, Shanghai Zhongshan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSY-LB-2014
Record Dates: First submitted 2014-04-17; First posted 2014-04-22 (Estimated); Last update posted 2016-06-13 (Estimated); Status verified 2016-06

CONDITIONS: Gastric and Esophageal Varices
Keywords: Gastric and Esophageal Varices; Hepatic Venous Pressure Gradient; Terlipressin; Octreotide
MeSH Terms: conditions — Esophageal and Gastric Varices | interventions — Terlipressin; Octreotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Terlipressin group (Experimental): Patients receive terlipressin 2 mg IV bolus
  Interventions: Drug: Terlipressin
- High Dose Octreotide group (Active Comparator): Patients receive Octreotide 50 μg/h with an initial bolus of 100 μg
  Interventions: Drug: Octreotide

INTERVENTIONS:
Drug: Terlipressin — Patients in the terlipressin group receive a single IV injection of 2 mg of terlipressin and a continuous IV infusion of normal saline.
  Other Names: HanWei
  Arms: Terlipressin group
Drug: Octreotide — Patients in high dose octreotide receive a single injection of 100μg octreotide and continuous IV infusion of 50 μg/h of octreotide.
  Other Names: ShanNing
  Arms: High Dose Octreotide group

SUMMARY:
The purpose of the study is to find patients's response to terlipressin and octreotide during hepatic venous pressure gradient measurement by observing portal and systemic hemodynamics.

DETAILED DESCRIPTION:
Esophageal variceal bleeding is one of the main causes of death in cirrhosis patients. Prevention of bleeding events, including primary and secondary prophylaxis, is very important for reducing the mortality of variceal bleeding. Terlipressin and octreotide can effectively control bleeding with few side effects, which has been recommended by Baveno V in treatment of acute variceal bleeding. Terlipressin and high dose octreotide will be administered to the patients with cirrhosis related esophageal varices when they undergo hepatic venous pressure gradient measurement. Changes from portal and systemic hemodynamics will be observed to evaluate the safety and effects of terlipressin and high dose octreotide as well as to determine wether patients respond to them. The results can be served as clinical evidence for preventing re-bleeding through long-acting terlipressin and octreotide in the future.

ELIGIBILITY:
Inclusion Criteria:

* Gastric and Esophageal Varices have been confirmed through endoscopy
* Liver Biopsy, CT or MRI indicates cirrhosis
* Patients who experienced variceal bleeding

Exclusion Criteria:

* The patients who are beyond the range from 18 to 80 years old
* The patients with unstable vital signs
* The patients with spontaneous peritonitis or other severe infections
* The patients with hepatorenal syndrome or renal inadequacy
* The patients with uncontrolled hepatic encephalopathy
* Pregnant and lactating women
* The patients who had contraindications for terlipressin or octreotide
* The patients who refuse to take part in this study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2014-02; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Fluctuation of HVPG | 10min, 20min and 30min after administration
  Terlipressin or octreotide will be administered to a patient once after the bottom line of his/her HVPG is determined. We observe the changes of HVPG after administration to find out the effects of terlipressin or octreotide on portal hemodynamics.

SECONDARY OUTCOMES:
Response Rate | 10min, 20min and 30min after administration
  Patients are considered responders when the HVPG decreases below 20 mmHg or by more than 10% from the baseline value

OTHER OUTCOMES:
Fluctuation of MAP and HR | 10min, 20min and 30min after administration
  Terlipressin or octreotide will be administered to a patient once after the bottom line of his/her mean arterial pressure and heart rate, as well as HVPG, are determined. We observe the changes of MAP and HR after administration to find out the effects of terlipressin or octreotide on systemic hemodynamics.
Incidence rate of complications | Participants will be followed for up to 24h starting from the moment of administration
  We intend to set incidence rate of complications associated with terlipressin or octreotide, to be specific, which include hypertension, abdominal pain, nausea, vomiting, diarrhea, headache, transient arrhythmia and vertigo. Participants will be followed for up to 24h starting from the moment of administration.

CONTACTS AND LOCATIONS:
Overall Officials: Shiyao Chen, Professor, Study Director — Shanghai Zhongshan Hospital
Locations (1):
- 180 Fenglin Road, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li B, Chen J, Zhang CQ, Wang GC, Hu JH, Luo JJ, Zhang W, Wei YC, Zeng XQ, Chen SY. The pharmacodynamic effect of terlipressin versus high-dose octreotide in reducing hepatic venous pressure gradient: a randomized controlled trial. Ann Transl Med. 2021 May;9(9):793. doi: 10.21037/atm-20-6774. PMID 34268406